CLINICAL TRIAL: NCT04790162
Title: Heartfulness Meditation to Improve Resilience Among Health Care Students: A 90 Day Program (HEART)
Brief Title: Heartfulness Meditation to Improve Resilience Among Health Care Students: A 90 Day Program
Acronym: HEART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-2951
Record Dates: First submitted 2021-03-04; First posted 2021-03-10 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Mental Health Wellness 1; Stress, Psychological; Depression; Anxiety
Keywords: Resiliency; Meditation; Health Care Student; Heartfulness
MeSH Terms: conditions — Stress, Psychological; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This is a randomized mixed methods (i.e., quantitative and qualitative methodology) intervention study with an experimental meditation group (HEART) and a wait-listed control group (CON). The wait-listed group will be offered the meditation after the 90-day data point.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meditation Intervention (Active Comparator): Heartfulness meditation
  Interventions: Behavioral: Heartfulness Meditation
- Control (No Intervention): Wait listed control group

INTERVENTIONS:
Behavioral: Heartfulness Meditation — Heartfulness meditation with a trainer provided virtually
  Arms: Meditation Intervention

SUMMARY:
This investigation will examine the feasibility of delivery and effect on resilience, depression and anxiety of a 90-day Heartfulness Practice delivered virtually for health care students. It is hypothesized that by providing this program on-line, students will be able to attend easily and complete the sessions. It is also hypothesized that those students who participate in the meditation program will increase resilience.

DETAILED DESCRIPTION:
This investigation will examine the feasibility of delivery and effect on resilience, depression and anxiety of a 90-day Heartfulness Practice delivered virtually for health care students.

SPECIFIC AIMS (SA) SA1: Determine feasibility and acceptability of delivering the 90-day Heartfulness Meditation Program virtually. Feasibility will be assessed by participant compliance, retention, and acceptability to the participants.

Criteria: Feasibility will be achieved by Compliance with average of at least 3 trainer led meditations / week Retention of 75% of participants at the end of 45 days (intermediate point) and 90 days (primary end point).

Criterion: Acceptability will be indicated by a CSQ8 score > 17. SA2: Examine the benefits of Heartfulness meditation on improving resilience, decreasing depression, and decreasing anxiety of health care students.

H2: At the end of 90 days (primary end point), students who participate in the Heartfulness Resilience Training (HEART) will have better resilience (CD-RISC) compared with students who do not participate and will have less anxiety and depression (HADS).

SA3: Examine the association between the number of sessions completed and changes in resilience, depression, and anxiety at 45 and 90 (primary end point) days.

H3: Changes in resilience, depression, and anxiety will be significantly correlated (Pearson correlation coefficients) with total number of sessions completed (H3a) and with number of one-on-one sessions with a trainer (H3b).

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 20-70
* Student in one of the health care programs on the Anschutz Medical Campus at the University of Colorado.

Exclusion Criteria:

* Students who are currently engaged in any formal meditation practice (e.g., Transcendental Meditation, Mindfulness Based Stress Reduction, (MBSR) more than once per week
* Unable to use the technology without special accommodations.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Feasibility as measured by the Number of Meditation Sessions Completed | 90 days
  Number of Meditation Sessions Completed-logged in RedCap
Change in Resilience as measured by Connor-Davidson Resilience Scale (CD-RISC) | Baseline, 45 days, 90 days
  25 item self-report questionnaire developed to quantify resilience and the impact of psychoeducation and resilience therapy techniques. Total scores range from 0-100 with higher scores indicating greater levels of resilience. The CD-RISC has been used in a variety of populations.
Change in Anxiety/Depression as measured by the Hospital Anxiety and Depression Scale (HADS) | Baseline, 45 days, 90 days
  14-item screening scale developed to indicate the potential presence of anxiety and depression. HADS consists of a 7-item anxiety subscale and a 7-item depression subscale. The HADS has good validity and reliability and has been studied in a variety of populations
Acceptability as measured by the Client Satisfaction Questionnaire (CSQ-8) | 45 days, 90 days
  8-item measure of satisfaction that is rated on a 4-point Likert scale and has a score range from 8 to 32. Higher scores indicate greater levels of satisfaction. For this study, we will assign 3 levels of satisfaction: 1) dissatisfied or least satisfied (score 8-16); 2) satisfied (score 17-30); and 3) very satisfied (score 31-32)The CSQ-8 has good test-retest reliability, internal consistency and sensitivity to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Robyn Gisbert, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No